CLINICAL TRIAL: NCT06779214
Title: Effect of Food-derived Active Components on Digestive Tract Health in Adults with Irritable Bowel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Xuyajun197673-03
Record Dates: First submitted 2024-11-24; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Syndrome - Diarrhoea
Keywords: Diarrhea-predominate Irritable bowel syndrome; probiotics; polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- resveratrol intervention (Experimental): participants receive different levels of resveratrol
  Interventions: Dietary Supplement: resveratrol_L; Dietary Supplement: resveratrol_H; Other: placebo_resveratrol
- prebiotic intervention (Experimental): subjects receive different levels of prebiotics
  Interventions: Dietary Supplement: Prebiotic_L; Dietary Supplement: Prebiotic_M; Dietary Supplement: Prebiotic_H; Other: placebo_Bif

INTERVENTIONS:
Dietary Supplement: Prebiotic_L — subject will receive a low-dosage (1*10^5) of Bifidobacterium. animalis subsp.Lactis A6 Strain
  Arms: prebiotic intervention
Dietary Supplement: resveratrol_L — subject will receive a low-dosage (300mg/d) of resveratrol
  Arms: resveratrol intervention
Dietary Supplement: Prebiotic_M — subject will receive a medium-dosage (1*10^8) of Bifidobacterium. animalis subsp.Lactis A6 Strain
  Arms: prebiotic intervention
Dietary Supplement: Prebiotic_H — subjects will receive a high-dosage (1*10^10) of Bifidobacterium. animalis subsp.Lactis A6 Strain
  Arms: prebiotic intervention
Dietary Supplement: resveratrol_H — subject will receive a low-dosage (600mg/d) of resveratrol
  Arms: resveratrol intervention
Other: placebo_Bif — subjects will receive placebo (one look-alike sunbstance that contains no prebiotics)
  Arms: prebiotic intervention
Other: placebo_resveratrol — subjects will receive placebo (one look-alike sunbstance that contains no resveratrol)
  Arms: resveratrol intervention

SUMMARY:
The goal of this clinical trial is to learn if Bifidobacterium. animalis subsp.

Lactis A6 Strain or resveratrol to improve the symptoms of diarrhea-predominate irritable bowel syndromes (IBS-D). The main questions it aims to answer are:

1. Does Bifidobacterium animalis subsp.Lactis A6 Strain or resveratrol improve the symptoms of IBS-D.
2. What is the optimal intervention dose of Bifidobacterium. animalis subsp.Lactis A6 Strain or resveratrol to improve IBS-D

Researchers will compare Bifidobacterium. animalis subsp.Lactis A6 Strain or resveratrol interventions to placebo (one look-alike sunbstance that contains no interventions substance) to see if Bifidobacterium. animalis subsp.Lactis A6 Strain or resveratrol relief the symptoms of patients with IBS-D.

Participants will:

1. Take Bifidobacterium. animalis subsp.Lactis A6 Strain or resveratrol every day for 30 days.
2. Visit the clinic once every 15 days for checkups and tests.

DETAILED DESCRIPTION:
We recruited patients with IBS-D. The subjects who met the inclusion criteria were randomly divided into placebo control group, Bifidobacterium. animalis subsp.Lactis A6 Strain group and resveratrol intervention. The intervention period lasted for 4 weeks, and the follow-up was conducted every 15 days. The main outcomes were: ① IBS Symptom Severity Scale (IBS-SSS), ② gut microbiota and their metabolites. The secondary outcomes were: ① IBS Quality of Life score (IBS-QOL), ② Bristol fecal traits score, ③hydrogen breath test; ④ Inflammatory markers. After the intervention, statistical analysis was performed on the experimental data to analyze and compare the differences in the main and secondary outcome indicators of the experimental groups, so as to clarify the intervention effect and effective intervention dose of probiotics and resveratrol on diarrheal IBS, and provide scientific basis for the formulation of relevant clinical treatment paths.

ELIGIBILITY:
Inclusion Criteria:

* met the Western Medicine Rome IV diagnostic criteria for diarrheal IBS
* 18 and 60 years old
* subjects voluntarily sign informed consent forms.

Exclusion Criteria:

* Having a disease that may affect the gut microbiome (e.g., inflammatory bowel disease, celiac disease, diabetes)
* Abdominal pain or diarrhea due to organic disease
* Patients with abdominal surgery
* Patients with serious mental illness and complications of heart, brain, liver, kidney and other systems
* Unable to communicate normally or skilled in the use of communication equipment
* Having serious mental problems or taking related drugs
* Drug or alcohol abusers
* People with special diets (such as vegetarians) or eating disorders or are receiving therapeutic dietary interventions
* Had used antibiotics, probiotics, other drugs that may affect the study
* Participants who are participating in other clinical trials
* Pregnant or lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Scale | 30 days
  it is a scale to evaluate the severity of irritable bowel syndrome symptoms, and the scoring range is from 0 to 500 points. The higher the score, the more severe the symptoms.
IBS Quality of Life | 30 days
  A scoring system is designed to mark changes in quality of life of patients, which includes 34 items with the score range of 34 to 170 scores. The higher the score, the poorer the quality of life.

SECONDARY OUTCOMES:
The levels of serum inflammatory cytokines, including interleukin-6 (IL-6), tumor necrosis factor-alpha (TNF-α), and interleukin-1β (IL-1β). | 30 days
  Using the ELISA method to detect inflammatory cytokines above mentioned in the serum of patients, higher levels of inflammatory cytokines suggest that the patient is in an inflammatory state.
Concentration of hydrogen in Hydrogen Breath Test | 30 days
  The hydrogen breath test is used to evaluate whether there is excessive overgrowth of small intestinal bacterial in patients. For subjects, the peak value of hydrogen exceeding 20ppm (parts per million) is considered positive, indicating the presence of small intestinal bacterial overgrowth.
the alpha diversity and composition of gut microbiome | 30 days
  16s rDNA is used to test the diversity and composition of gut microbiome of participants. The alpha diversity is adopted to evaluate the number of species within a community (richness) as well as the distribution of each species (evenness). the higher the indicator, the healthier the gut. The composition of gut microbiome is used to describe the abundance of beneficial and harmful bacteria. The higher the abundance of beneficial bacteria and the lower the abundance of harmful bacteria, the healthier the gut is.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No